CLINICAL TRIAL: NCT04371367
Title: A Double-blind, Randomized Study Versus Placebo of Avdoralimab (IPH5401), an Anti-C5aR Antibody, in Patients With COVID-19 Severe Pneumonia
Brief Title: Avdoralimab an Anti-C5aR Antibody, in Patients With COVID-19 Severe Pneumonia ( FORCE )
Acronym: FORCE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Collaborators: Innate Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-21
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: COVID
MeSH Terms: interventions — avdoralimab

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- avdoralimab (Experimental): Biological/Vaccine: avdoralimab intravenous administration of avdoralimab
  Other Names:
  • IPH5401
  Interventions: Biological: avdoralimab
- Placebo (Placebo Comparator): intravenous administration of Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: avdoralimab — intravenous administration of avdoralimab
  Other Names: IPH5401
  Arms: avdoralimab
Other: Placebo — intravenous administration of placebo
  Arms: Placebo

SUMMARY:
The primary objective of this trial is to improve the proportion of COVID-19 patients with severe pneumonia who no longer need to be hospitalized, and to reduce the need for and duration of mechanical ventilation in patients with COVID-19 pneumonia complicated by acute respiratory distress syndrome (ARDS).

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 severe pneumonia patients need for oxygen therapy ≥ 5 l/min or high-flow oxygen therapy
* COVID-19 related Acute Respiratory Distress Syndrome (ARDS) requiring mechanical ventilation

Exclusion Criteria:

* Pregnant woman
* Uncontrolled sepsis of bacterial or fungal origin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Clinical improvement using WHO ordinal scale | day 28
  improvement of WHO ordinal scale
Number of ventilator-free days at Day 28 (VFD28) | day 28
  Number of days without mechanical ventilation at Day 28 for COVID-19 related Acute Respiratory Distress Syndrome (ARDS) Patients hospitalized in ICU

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | day 28

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Garrido-Pradalie, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carvelli J, Meziani F, Dellamonica J, Cordier PY, Allardet-Servent J, Fraisse M, Velly L, Barbar SD, Lehingue S, Guervilly C, Desgrouas M, Camou F, Piperoglou C, Vely F, Demaria O, Karakunnel J, Fares J, Batista L, Rotolo F, Viotti J, Boyer-Chammard A, Lacombe K, Le Dault E, Carles M, Schleinitz N, Vivier E; FOR COVID Elimination (FORCE) Study Group. Avdoralimab (Anti-C5aR1 mAb) Versus Placebo in Patients With Severe COVID-19: Results From a Randomized Controlled Trial (FOR COVID Elimination [FORCE]). Crit Care Med. 2022 Dec 1;50(12):1788-1798. doi: 10.1097/CCM.0000000000005683. Epub 2022 Oct 10. PMID 36218354
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343